CLINICAL TRIAL: NCT02150863
Title: Treatment of Field Cancerization for Reduction in Tumor Burden - A Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling participants due to exclusion and inclusion criteria
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Harvard Medical School Professor in dermatology, Director of the Wellman Center for Photomedicine; and adjunct Professor of Health Sciences and Technology at MIT, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P000121
Record Dates: First submitted 2014-03-10; First posted 2014-05-30 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Extensive Photodamage; Actinic Keratosis; History of Numerous Skin Cancers
Keywords: actinic keratosis; field cancerization; organ transplant patients
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ultrapulse laser alone (Active Comparator)
  Interventions: Device: Ultrapulse Carbon Dioxide Laser
- Ultrapulse laser plus Cellutome Harvesting system (Active Comparator)
  Interventions: Device: Ultrapulse Carbon Dioxide Laser; Device: Cellutome epidermal harvesting system
- Control (No Intervention)

INTERVENTIONS:
Device: Ultrapulse Carbon Dioxide Laser
  Other Names: Lumenis Ultrapulse
  Arms: Ultrapulse laser alone; Ultrapulse laser plus Cellutome Harvesting system
Device: Cellutome epidermal harvesting system
  Arms: Ultrapulse laser plus Cellutome Harvesting system

SUMMARY:
This project aims to treat field cancerization ( pre-skin cancers) in a manner that will reduce the future pre-skin cancers and non-melanoma skin cancers in patients with significant photodamage.

This is 3 year prospective, randomized, controlled comparison of a single treatment with carbon dioxide laser resurfacing vs. carbon dioxide resurfacing plus autologous epidermal skin graft from a non sun exposed site vs. control.

Thirty subjects will receive treatment with each of the modalities.

The primary measures of efficacy are (a) count of the number of actinic keratosis and non melanoma skin cancers, (b) blinded evaluation of severity from standard digital photographs taken before and after the treatments, and (c) change in histology before and after treatment. Safety measures include (a) pain, (b) scarring, (c) wound healing, (d) and infection

ELIGIBILITY:
Inclusion criteria

1. Subjects with ages between 18 and 85 years, male or female.
2. Subjects with at least 4 clinically diagnosed actinic keratoses (AKs) per treatment site ( up to 200 sq cm), excluding the face and neck
3. Subjects with history of at least 1 non-melanoma skin cancer within the past year
4. Willingness to participate in the study
5. Informed consent agreement signed by the subject
6. Willingness to follow the treatment schedule and post treatment care requirements
7. Willingness to not use topical or systemic (oral) TREATMENT medications including imiquimod, 5-Fluorouracil, photodynamic therapy, during the treatment period.
8. Has not had treatment for AKs in the treatment area for 4 weeks prior to enrollment

Exclusion criteria

1. Subjects with active skin cancer in the treatment area. Once the non-melanoma skin cancer has been treated, the subject can be immediately enrolled.
2. Infection of the area to be treated
3. An open wound in the area to be treated
4. Presence of suntan in the area to be treated, or active tanning during the study
5. Subjects who have taken medication known to induce photosensitivity in the previous 3 months
6. The patient has any contraindication to use of the carbon dioxide laser, including but not limited to, intake of isotretinoin in past 12 months; patients with reduced adnexal structures (eg, scleroderma, irradiation or burns); patients with history of vitiligo or psoriasis (risk of Koebnerization); history of keloids/hypertrophic scarring.
7. Subject is unable to comply with treatment, home care or follow-up visits
8. Subject is pregnant or breast feeding
9. Prior use of topical retinoids, 5 fluorouracil, or imiquimod in treated areas within one month of initial treatment
10. Prior skin treatment with laser or other devices in the treated area within two months of initial treatment or during the course of the study;
11. Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
12. Concurrent inflammatory skin conditions, including, but not limited to, eczema, contact dermatitis of any severity;
13. Active Herpes Simplex at the time of treatment;
14. Multiple dysplastic nevi in area to be treated;
15. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to each treatment (as per the patient's physician discretion);
16. Significant concurrent illness, such as uncontrolled diabetes, (i.e., any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process);
17. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
18. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or study personnel) to treat the subject as part of this research study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rox Anderson, MD, Principal Investigator — Massachusetts General Hospital/ Wellman Center for Photomedicine
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrapulse Laser Alone: Ultrapulse Carbon Dioxide Laser
- Ultrapulse Laser Plus Cellutome Harvesting System: Ultrapulse Carbon Dioxide Laser
  Cellutome epidermal harvesting system
- Control: Control group, no treatment
Period: Overall Study
Arm/Group | Ultrapulse Laser Alone | Ultrapulse Laser Plus Cellutome Harvesting System | Control
Started | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There was only one patient enrolled in this study
Groups:
- Control: Control group
- Total: Total of all reporting groups
Arm/Group | Ultrapulse Laser Alone | Ultrapulse Laser Plus Cellutome Harvesting System | Control | Total
Number analyzed (Participants) | 0 | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 0 | 0 |  | 0
  >=65 years | 0 | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 70 |  | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 |  | 1
  Male |  | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 0
  Not Hispanic or Latino |  | 1 |  | 1
  Unknown or Not Reported |  | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Count of the Number of Actinic Keratosis and Non Melanoma Skin Cancers in the Treatment Area
Description: This is done at every visit over the 3 year period
Time Frame: Entire study period (3 years)
Population: Zero participants were analyzed because no patients finished this study. Patient recruitment was very difficult for this study, and therefore the study ended prematurely.
Groups:
- Control: Control group (no laser or CelluTome)
Arm/Group | Ultrapulse Laser Alone | Ultrapulse Laser Plus Cellutome Harvesting System | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The time the patient was in the study, 6 months
Description: For areas where participants at risk is 0, it is because there were no participants in these categories.
Groups:
- Control: Control site
Arm/Group | Ultrapulse Laser Alone | Ultrapulse Laser Plus Cellutome Harvesting System | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Recruitment was very difficult for this study. Due to long study period, patient retention was also difficult. The study was terminated because of low recruitment. One subject started the study and was lost to follow-up, without completing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-12-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02150863/Prot_000.pdf